CLINICAL TRIAL: NCT06396559
Title: Development of the Orientation Training Mobile Support Application and Its Effect on the Anxiety Level and Patient Safety Attitude Of Student Nurses: Pre Test After Test Randomized Controlled Study
Brief Title: Orientation Training Mobile Support Application for Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Ezgi Yorgancılar, principal investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nec Erbakan Uni Health Science
Record Dates: First submitted 2023-12-21; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Nurse-Patient Relations
Keywords: student nurse; mobile application; patient safety; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (No Intervention): Student nurses will undertake internships included in their curriculum.
- mobil application (Experimental): Student nurses will undertake internships included in their curriculum. They will use the patient safety mobile application during the internship.
  Interventions: Behavioral: pre test-post test

INTERVENTIONS:
Behavioral: pre test-post test — The mobile application will be installed on the mobile devices of student nurses and its effectiveness will be tested.
  Other Names: mobile application
  Arms: mobil application

SUMMARY:
Mobile health (mHealth) applications are shifting mobile phone technology from the simple function of text messaging to a dynamic, interactive, and social environment that includes verbal, audio, and visual messages. The widespread adoption of mobile phones and smartphones offers a promising opportunity for health promotion. The use of modern mobile technology (phone calls and texts, videos, internet and smartphone applications) is becoming increasingly popular in the healthcare field and is used to inform and guide patients in a variety of chronic diseases. The number of mobile phone subscribers worldwide is approximately five billion. In low- and middle-income countries, the spread of mobile phones is occurring faster than other infrastructure developments. In low- and middle-income countries, mobile information technology interventions are considered complementary approaches to deliver health-related information.

In line with the contemporary education approach, nursing students' clinical stress and anxiety must be taken under control by making student-centered arrangements in education, strengthening students' perception of the profession, and creating appropriate learning environments. It is important to adapt mobile support application models compatible with the national health system at institutional and national levels in the planning of education and training due to reasons such as the excitement, anxiety and fear that students feel before clinical practice, and the inadequacy in the number of instructors and nurses. Clinical stress and anxiety of nursing students should be taken under control by making student-centered arrangements in education in line with the contemporary education approach, strengthening students' perception of the profession, and creating appropriate learning environments. It is important to adapt mobile support application models compatible with the national health system at institutional and national levels in the planning of education and training due to reasons such as the excitement, anxiety and fear that students feel before clinical practice, and the inadequacy in the number of instructors and nurses.

DETAILED DESCRIPTION:
Mobile health (mHealth) applications are shifting mobile phone technology from the simple function of text messaging to a dynamic, interactive, and social environment that includes verbal, audio, and visual messages. The widespread adoption of mobile phones and smartphones offers a promising opportunity for health promotion. The use of modern mobile technology (phone calls and texts, videos, internet and smartphone applications) is becoming increasingly popular in the healthcare field and is used to inform and guide patients in a variety of chronic diseases. The number of mobile phone subscribers worldwide is approximately five billion. In low- and middle-income countries, the spread of mobile phones is occurring faster than other infrastructure developments. In low- and middle-income countries, mobile information technology interventions are considered complementary approaches to deliver health-related information.

In line with the contemporary education approach, nursing students' clinical stress and anxiety must be taken under control by making student-centered arrangements in education, strengthening students' perception of the profession, and creating appropriate learning environments. It is important to adapt mobile support application models compatible with the national health system at institutional and national levels in the planning of education and training due to reasons such as the excitement, anxiety and fear that students feel before clinical practice, and the inadequacy in the number of instructors and nurses. Clinical stress and anxiety of nursing students should be taken under control by making student-centered arrangements in education in line with the contemporary education approach, strengthening students' perception of the profession, and creating appropriate learning environments. It is important to adapt mobile support application models compatible with the national health system at institutional and national levels in the planning of education and training due to reasons such as the excitement, anxiety and fear that students feel before clinical practice, and the inadequacy in the number of instructors and nurses.

.

ELIGIBILITY:
Inclusion Criteria:

* Being a fourth year student at the Faculty of Nursing.
* Taking the vocational practice course.
* Owning a smartphone with Android or iOS operating system.
* Being able to speak and understand Turkish.

Exclusion Criteria:

* Not being a fourth-year student of the faculty of nursing.
* Not taking the professional practice course.
* Not owning a smartphone with Android or iOS operating system.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Development of the Orientation Training Mobile Support Application and Its Effect on the Anxiety Level and Patient Safety Attitude Of Student Nurses: Pre Test After Test Randomized Controlled Study | After 1 month and 3 month, student nurses' patient safety attitude scores will be measured.
  Orientation Training Mobile Support Application

IPD SHARING:
Plan to Share IPD: No
Since this mobile application for patient safety will be developed by the researcher, it will not be made available to other researchers.

REFERENCES:
- [Background] O'Connor S, Andrews T. Mobile technology and its use in clinical nursing education: a literature review. J Nurs Educ. 2015 Mar;54(3):137-44. doi: 10.3928/01484834-20150218-01. Epub 2015 Feb 19. PMID 25693246